CLINICAL TRIAL: NCT04883840
Title: Drug Repurposing - Statins as Microbiota Modulating Agents in Ulcerative Colitis
Acronym: ReMiDy
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to the university's termination of its contract with the online questionnaire platform, we decided to discontinue the study before reaching the anticipated sample size.
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Vlaams Instituut Biotechnologie (VIB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: S63190
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Ulcerative Colitis
Keywords: Microbiome; Dysbiosis
MeSH Terms: conditions — Colitis, Ulcerative; Dysbiosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Rosuvastatin 10mg
- Rosuvastatin 10 mg (Experimental)
  Interventions: Drug: Rosuvastatin 10mg

INTERVENTIONS:
Drug: Rosuvastatin 10mg — Daily dose of one medication over 8 week period then switch to another medication over an 8 week period (type of medication during each intervention period is blinded and then randomized).

SUMMARY:
* Evaluation of the microbiota modulation away from inflammation associated microbiota profile Bacteroides2 (Bact2)
* Evaluation of the effect of microbiota modulation on disease activity in ulcerative colitis and Crohn's disease patients.

ELIGIBILITY:
Inclusion criteria

General criteria Willingness to participate in the study and to sign the informed consent (Dutch) Between 18 and 70 years old Access to a -20°C freezer

Criteria specific to UC patients In clinical remission (total Mayo Score below 4) or with currently mild to moderate active ulcerative colitis (Mayo Score between 4-10 and endoscopic sub score 2-3 at week 0), either untreated or under stable medication

Criteria specific to CD patients In clinical remission (CDAI score below 150 at week 0) or with currently mild active Crohn's disease (CDAI score between 150-220 at week 0), either untreated or under stable medication

Exclusion criteria

General criteria Prior and/or ongoing use of statins Females who are pregnant, actively trying to become pregnant, or are not using effective anticonception measures Active liver disease or liver damage including unexplained persistent elevations of serum transaminases and any serum transaminases elevation exceeding three times the upper limit of normal (ULN) Prediabetes Personal or family history of or diagnosed with hereditary muscular disorders History of or diagnosed with alcohol abuse Use of antibiotics at any time in the four weeks before the start of the intervention (UC & CD patients Participation in simultaneously occurring clinical trials

Criteria specific to CD & UC patients Any surgical intervention in the gastrointestinal tract (with the exception of an appendectomy in all participants or ileocecal resections, cholecystectomy, fistulectomy, strictureplasty and abscess drainage in CD patients.) Severe renal impairment (creatinine clearance <30 ml/min) Diabetes mellitus Hypothyroidism Myopathy Other conditions leading to profound immunosuppression such as HIV, infectious diseases, bone marrow malignancies, and liver cirrhosis Use of methotrexate or calcineurin inhibitors Indeterminate colitis Steroid dependency, i.e., requiring more than 16mg Medrol (methyl prednisone) or an equivalent steroid two weeks before week 0

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2020-10-22 (Actual); Primary Completion 2025-10-11 (Actual); Study Completion 2025-10-11 (Actual)

PRIMARY OUTCOMES:
Significant change in gastrointestinal microbiome composition | 8 weeks
  Change away from dysbiotic enterotype to eubiotic one when taking IMP

SECONDARY OUTCOMES:
UC Mayo Score / CDAI | 8 weeks
  Significant improvement in UC patient overall disease status characterised by reduction of at least 3 points in the non-invasive Mayo Score and by a full point reduction in the endoscopic subscore. Similarly, significant improvement in CD patient overall disease status characterised by reduction of the Crohn's disease activity index (CDAI) by at least 70 points or by a CDAI score < 150

CONTACTS AND LOCATIONS:
Overall Officials: Severine Vermeire, MD & PhD, Principal Investigator — KU/UZ Leuven; Jeroen Raes, PhD, Study Director — KU Leuven/VIB
Locations (3):
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden, Antwerp
  - UZ Leuven, Leuven, Vlaams-Brabant
  - AZ Delta, Roeselare, West-Vlaanderen

IPD SHARING:
Plan to Share IPD: Undecided